CLINICAL TRIAL: NCT04526795
Title: Phase Ib Study of Fludarabine, Cytarabine (Ara-C) and Pegylated Erwinase (Pegcrisantaspase) in Patients with Relapsed or Refractory Leukemia
Brief Title: Fludarabine, Cytarabine, and Pegcrisantaspase for the Treament of Relapsed or Refractory Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administratively Complete
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0434; NCI-2020-05459 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0434 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-08-13; First posted 2020-08-26 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Blast Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Recurrent Acute Biphenotypic Leukemia; Recurrent Acute Lymphoblastic Leukemia; Recurrent Acute Myeloid Leukemia; Recurrent Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Recurrent T-Cell Prolymphocytic Leukemia; Refractory Acute Biphenotypic Leukemia; Refractory Acute Lymphoblastic Leukemia; Refractory Acute Myeloid Leukemia; Refractory Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Refractory T-Cell Prolymphocytic Leukemia
MeSH Terms: conditions — Blast Crisis; Leukemia, Biphenotypic, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Prolymphocytic, T-Cell | interventions — Cytarabine; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pegcrisantaspase, fludarabine, cytarabine) (Experimental): INDUCTION: Patients receive pegcrisantaspase IV over 60 minutes on days 1 and 15, and fludarabine IV over 15-30 minutes and cytarabine IV over 2 hours on days 8-11 in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients receive pegcrisantaspase IV over 60 minutes on days 1 and 15, and fludarabine IV over 15-30 minutes and cytarabine IV over 2 hours on days 8-10. Treatment repeats every 5 weeks for up 3 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cytarabine; Drug: Fludarabine; Drug: Pegcrisantaspase

INTERVENTIONS:
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Drug: Pegcrisantaspase — Given IV

SUMMARY:
This phase Ib trial investigates the side effects and best dose of pegcrisantaspase when given together with fludarabine and cytarabine for the treatment of patients with leukemia that has come back (relapsed) or has not responded to treatment (refractory). Pegcrisantaspase may block the growth of cancer cells. Chemotherapy drugs, such as fludarabine and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving pegcrisantaspase in combination with fludarabine and cytarabine may work better in treating patients with leukemia compared to the combination of fludarabine and cytarabine.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety and tolerability of fludarabine, cytarabine (araC), and pegcrisantaspase in patients with relapsed and refractory leukemias.

SECONDARY OBJECTIVES:

I. To determine the overall response rate (complete remission [CR], CR with incomplete count recovery [CRi], partial remission [PR], or morphologic leukemia free state [MLFS]) of a lead-in dose of single-agent pegcrisantaspase in patients with relapsed and refractory leukemias.

II. To determine the overall response rate (complete remission [CR], CR with incomplete count recovery [CRi], partial remission [PR], or morphologic leukemia free state [MLFS]) of fludarabine, araC, and pegcrisantaspase in patients with relapsed and refractory leukemias.

III. To assess overall survival (OS) and disease-free survival (DFS) of patients treated with fludarabine, araC, and pegcrisantaspase.

IV. To assess the duration of response to the combination in patients with advanced leukemias.

V. To characterize the pharmacokinetics (PK) pharmacodynamics (PD) anti-drug antibodies (ADA) of pegcrisantaspase in patients with relapsed and refractory leukemias.

EXPLORATORY OBJECTIVE:

I. Explore pretreatment and on-treatment biological correlates to predict sensitivity/resistance of pegcrisantaspase-based therapy.

OUTLINE: This is a dose-escalation study of pegcrisantaspase.

INDUCTION: Patients receive pegcrisantaspase intravenously (IV) over 60 minutes on days 1 and 15, and fludarabine IV over 15-30 minutes and cytarabine IV over 2 hours on days 8-11 in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION: Patients receive pegcrisantaspase IV over 60 minutes on days 1 and 15, and fludarabine IV over 15-30 minutes and cytarabine IV over 2 hours on days 8-10. Treatment repeats every 5 weeks for up 3 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of relapsed or refractory leukemia including, but not limited to acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), T-cell prolymphocytic leukemia, biphenotypic acute leukemia, or blast-phase of chronic myeloid Leukemia (CML) will be allowed during the safety lead-in phase
* For cohort A of the expansion phase: Patients with a diagnosis untreated adverse-risk AML (as defined by ELN [European Leukemia Net Classification] 2017) will be enrolled
* For cohort B of the expansion phase: Patients with a diagnosis of relapsed or refractory AML will be enrolled
* Bilirubin =< 2 mg/dL
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN)
* Creatinine =< 1.5 x ULN
* Cardiac ejection fraction of > or = 45% within the past 3 months
* Amylase and lipase =< 1.5 x ULN
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* A negative urine pregnancy test is required within one week (7 days) for all women of childbearing potential prior to being registered on this trial
* Patient must have the ability to understand the requirements of the study and signed informed consent. A signed informed consent by the patient or his legally authorized representative is required prior to their enrollment on the protocol

Exclusion Criteria:

* Pregnant women are excluded from this study because the agents used in this study have the potential for teratogenic or abortifacient effects. Because there is a potential risk for adverse events in nursing infants secondary to treatment of the mother with the chemotherapy agents, breastfeeding should also be avoided
* Uncontrolled intercurrent illness including, but not limited to active uncontrolled infection, symptomatic congestive heart failure (New York Heart Association [NYHA] class III or IV), unstable angina pectoris, clinically significant cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patient with documented hypersensitivity to any of the components of the chemotherapy program
* Prior treatment with pegylated asparaginase
* Patients with a diagnoses of acute promyelocytic leukemia (AML-M3) will be excluded from this trial
* Men and women of childbearing potential who do not practice contraception. Women of childbearing potential and men must agree to use contraception prior to study entry and for the duration of study participation. Effective methods of birth control include:

  * Birth control pills, shots, implants or patches
  * Intrauterine devices (IUDs)
  * Condom or occlusive cap (diaphragm or cervical/vault caps) used with spermicide
  * Abstinence
  * Females of non-childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation, oophorectomy, and/or hysterectomy
* Patients with history of clinically significant venous thromboembolism

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | End of cycle 1 (5 weeks)
  Measured by dose limiting toxicities (DLTs). DLTs will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE, version 5) by organ system. DLT will be defined as drug-related adverse events during cycle one (during the lead-in phase).

SECONDARY OUTCOMES:
Overall response rate (ORR) of pegcrisantaspase | Up to 20 weeks
  The overall response rate for each cohort will be calculated and confidence interval will be provided. Chi square test or Fisher's exact test will be used to evaluate the association between patient prognostic factor and response.
ORR of fludarabine, cytarabine (araC), and pegcrisantaspase | Up to 20 weeks
  The overall response rate for each cohort will be calculated and confidence interval will be provided. Chi square test or Fisher's exact test will be used to evaluate the association between patient prognostic factor and response.
Overall survival (OS) | From date of treatment start until date of death due to any cause, assessed up to 20 weeks
  Will be estimated using the method of Kaplan and Meier. Comparison of time-to-event endpoints by important subgroups will be made using the log-rank test.
Disease-free survival (DFS) | From date of remission until the date of first objective documentation ofdisease-relapse or death, assessed up to 20 weeks
  Will be estimated using the method of Kaplan and Meier. Comparison of time-to-event endpoints by important subgroups will be made using the log-rank test.
Duration of response | Up to 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tapan M Kadia, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org